CLINICAL TRIAL: NCT04512950
Title: Crystalloid FLUID Choices for Resuscitation of Hospital Patients: A Pragmatic Cluster Cross Over Trial
Brief Title: Crystalloid FLUID Choices for Resuscitation of Hospitalized Patients
Acronym: FLUID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0778
Record Dates: First submitted 2019-06-03; First posted 2020-08-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Fluid Therapy
Keywords: Ringer's Lactate; 0.9% saline; Resuscitation; Hypovolemia; Rehydration
MeSH Terms: conditions — Hypovolemia | interventions — Ringer's Lactate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Cluster Cross Over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ringer's lactate (Active Comparator): administered as infusions or boluses as per the treating physician
  Interventions: Drug: Ringer's lactate
- 0.9% Saline (Active Comparator): administered as infusions or boluses as per the treating physician
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Ringer's lactate — Half of the hospitals will be randomized to Ringer's Lactate for a 12 week study period; after a 2 week run-out, the study fluid will be switched to 0.9% saline for another 12 week study period, followed by a 2 week run-out.
  Other Names: Lactated Ringer's
  Arms: Ringer's lactate
Drug: 0.9% saline — Half of the hospitals will be randomized to 0.9% saline for a 12 week study period; after a 2 week run-out, the study fluid will be switched to Ringer's Lactate for another 12 week study period, followed by a 2 week run-out.
  Other Names: sodium chloride 0.9%
  Arms: 0.9% Saline

SUMMARY:
The aim of the FLUID Trial is to conduct a pragmatic, multi-centre, open label randomized cluster cross-over trial (RCT) to determine whether fluid administration with 0.9% saline as compared to Ringer's lactate decreases death or re-admission to hospital with 90 days of the index admission.

DETAILED DESCRIPTION:
Crystalloid fluids are used extensively for acutely ill patients who are admitted to hospital. Two fluids most commonly used are 0.9% saline and Ringer's Lactate. Both are used to rehydrate patients, restore fluid volume and help stabilize blood pressure and failing organ and both have been used for several decades. Until recently, it was thought the fluids are essentially equivalent other than some minor differences related to the concentration of salt components (sodium and chloride) and buffers (Ringer's Lactate has lactate as a buffer). The safety of 0.9% saline is now being questioned due to its high chloride content and its association with the development of hyperchloremic metabolic acidosis. Until recently, the evidence base supporting the superiority of Ringer's Lactate has been derived from observational studies. Two recent pilot studies in critically ill patients comparing 0.9% saline to balanced crystalloid fluids (Ringer's lactate and/or Plasma-Lyte, another balanced crystalloid) did not detect clinical outcome differences between the fluid groups, but the trials were not powered to do so. Furthermore, two multiple period cluster cross-over studies conducted at one institution comparing 0.9% saline to balanced crystalloids (Ringer's lactate and Plasma-Lyte) in the emergency department (ED) and intensive care unit (ICU) found small differences in a composite outcome which included death, requirement for dialysis or persistent renal dysfunction, in favor of balanced crystalloids. In contrast, two large multi-centre randomized trials (BaSICS, n=11 052 and PLUS, n=5037) examined the efficacy of NS as compared with a balanced crystalloid (RL and Plasma-Lyte 148, respectively) on the primary outcome 90-day mortality. Neither of these trials detected a difference in 90-day mortality; in BaSICS, the mortality rate was 22.0% versus 21.8%; in PLUS, mortality was 27.2% versus 26.4%. Renal function did not differ between the fluid groups in either trial, although the PLUS trial was stopped early due to recruitment challenges and insufficient funding during the pandemic. In a systematic review of 13 critical care trials to January 2022 and 35 884 participants, there were no detectable differences in renal function. In low risk of bias trials, there was no significant difference in mortality for the 0.9% saline as compared with balanced crystalloid group (28.2% and 27.9%, respectively; relative risk (RR) 0.96 (95% CI 0.91 to 1.01)), nor renal function. However, authors concluded that there is a high probability balanced crystalloids reduce death since the CIs ranged from a 9% relative reduction to a 1% relative increase in death. Authors and editorialists urge the conduct of large multi-centre randomized trials, with longer-term patient centred outcomes supported by health economic evaluations to provide confirmatory evidence to guide future clinical practice and resource allocation related to these usual care crystalloid fluids.

Small differences in clinical outcomes between crystalloid resuscitation fluids are highly relevant. Furthermore, small absolute differences in important clinical outcomes may translate into substantial savings to hospitals and the health care system. The FLUID trial will determine if there are differences in the clinically important outcomes of death and hospital re-admissions. FLUID is novel in its design because it is a hospital wide pragmatic cluster cross-over comparative effectiveness trial that will be conducted in both academic and community sites which will use provincial health administrative data available through the Institute of Clinical Evaluative Sciences (ICES) for all clinical data collection. Our trial will answer this fundamental fluid resuscitation question and determine if Ringer's Lactate is superior to 0.9% saline at much lower cost in comparison to an individual patient randomized controlled trial (RCT), or even a conventional cluster RCT.

ELIGIBILITY:
Inclusion Criteria:

● All adult and pediatric patients with an index admission to the participating hospitals during study periods

Exclusion Criteria:

* neonates
* physicians may opt out of the use of the allocated study fluid for a specific patient

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43626 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-13 (Actual)

PRIMARY OUTCOMES:
Number of participants that died or were readmitted to hospital | 90 days from index hospital admission
  the number of deaths or readmission to hospital

SECONDARY OUTCOMES:
Number of participants that died | 90 days from index hospital admission
  The number of deaths
Number of participants re-admitted to hospital | 90 days from index hospital admission
  the number of participants re-admitted to any hospital in Ontario
Number of participants that required dialysis or continuous renal replacement therapy | 90 days from index hospital admission
  the number of participants who required the initiation of dialysis or continuous renal
  replacement therapy in the first 90 days from index hospital admission with no history of renal disease requiring dialysis in the previous 6 months
Number of participants that required re-intubation in the post anesthetic care unit operative period | Up to 90 days after the initial operation during index hospital admission
  the number of post operative participants who failed their initial extubation and required re-intubation in the post anesthetic care unit within 1 day of their initial surgery during index hospital admission
Duration of hospitalization | Up to 90 Days from index hospital admission
  the number of days participants were hospitalized during index admission
ED visits | number of index ED visits within 90 days of index hospital admission
  number of index ED visits
Discharged to a facility other than home | 90 days from index hospital admission
  number of participants discharged from index hospitalization to a facility other than home
Number of patients that required a re-operation | Up to 90 days after the initial operation during index hospital admission
  Number of patients that required a re-operation after an initial surgery during index hospital admission surgery during the index hospitalization

OTHER OUTCOMES:
Incremental cost, life-year saved, quality-adjusted life-year (QALY) | 90 days from index hospitalization
  cost per life-year saved and cost per QALY gained

CONTACTS AND LOCATIONS:
Overall Officials: Lauralyn McIntyre, MS MHSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (7):
- Canada (7):
  - Hamilton General Hospital, Hamilton, Ontario
  - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Montfort Hospital, Ottawa, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - The Ottawa Hospital Civic Campus, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
all data will be obtained from the Institute of Clinical Evaluative Sciences - no individual patient data will be obtained

REFERENCES:
- [Derived] McIntyre L, Fergusson D, McArdle T, English S, Cook DJ, Fox-Robichaud AE, Martin C, Marshall J, Pugliese M, Menon K, Thavorn K, Graham ID, Hawken S, Iyengar A, Kyeremanteng K, Saginur R, Seely AJE, Stiell IG, Bainbridge D, Weijer C, Taljaard M; Canadian Critical Care Trials Group. A Crossover Trial of Hospital-Wide Lactated Ringer's Solution versus Normal Saline. N Engl J Med. 2025 Aug 14;393(7):660-670. doi: 10.1056/NEJMoa2416761. Epub 2025 Jun 12. PMID 40503714
- [Derived] Shaw JF, Ouyang Y, Fergusson DA, McArdle T, Martin C, Cook D, Graham ID, Hawken S, McCartney CJL, Menon K, Saginur R, Seely A, Stiell I, Fox-Robichaud A, English S, Marshall J, Thavorn K, Taljaard M, McIntyre LA; Canadian Critical Care Trials Group. A Hospital-Wide Open-Label Cluster Crossover Pragmatic Comparative Effectiveness Randomized Trial Comparing Normal Saline to Ringer's Lactate: Protocol and Statistical Analysis Plan of The FLUID Trial. JMIR Res Protoc. 2023 Oct 6;12:e51783. doi: 10.2196/51783. PMID 37801356